CLINICAL TRIAL: NCT06849505
Title: Closed - Loop Neuromodulation of Post - Stroke Motor Dysfunction by Transcranial Magnetic Stimulation Synchronized with Specific Motor Task Training
Brief Title: Transcranial Magnetic Stimulation Synchronized with Motor Task Training for Post-Stroke Rehabilitation
Acronym: TMS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital of the Chinese People's Liberation Army Naval Medical University (Other)
Collaborators: shanghai center for brain science and brain-inspired technology (Unknown)
Responsible Party: Principal Investigator, Xiaonan Huang, Principal Investigator, First Affiliated Hospital of the Chinese People's Liberation Army Naval Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CHEC2025-055
Record Dates: First submitted 2025-02-19; First posted 2025-02-27 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Stroke; Upper Extremity Parasis
Keywords: stroke; individualized; TMS; motor dysfunction; online
MeSH Terms: conditions — Stroke; Neurologic Manifestations

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- online rTMS (Experimental): In the online stimulation group, the TMS treatment will continuously adjust the TMS parameters according to the baseline data and the data changes during the treatment to achieve personalized intervention. When patients receive TMS treatment, it is combined with upper limb movement tasks. When the task starts autonomously, TMS stimulation is triggered through electromyographic feedback. When the task stops or is completed, the TMS stimulation also stops immediately according to the electromyographic feedback, achieving real - time effects.
  Interventions: Device: online rTMS
- offline rTMS (Active Comparator): For the offline stimulation group, TMS treatment will be carried out before the task starts. After the stimulation ends, the subjects will then complete the task.
  Interventions: Device: offline rTMS
- sham rTMS (Sham Comparator): Patients in the sham group also receive sham stimulation treatment combined with specific tasks, which is the same as the online stimulation group, except that the TMS stimulation is sham stimulation.
  Interventions: Device: sham rTMS

INTERVENTIONS:
Device: online rTMS — 5 Hz rTMS is applied to the MRI-localized hotspot on the affected hemisphere when the patients are performing motor tasks
  Arms: online rTMS
Device: offline rTMS — The patients perform motor tasks after 5 Hz rTMS applied to the MRI-guided hotspot on the affected hemisphere
  Arms: offline rTMS
Device: sham rTMS — Sham rTMS is applied to the M1 on the affected hemisphere when the patients are performing motor tasks.
  Arms: sham rTMS

SUMMARY:
The goal of this clinical trials is to investigate the effectiveness of individualized online repetitive transcranial magnetic stimulation (rTMS) in enhancing upper limb motor rehabilitation during the subacute and chronic phase of stroke. It will also learn about the safety of individualized online rTMS intervention methods. The main questions it aims to answer are:

Does rTMS synchronized with motor training improve motor rehabilitation in patients with the ability to induce motor evoked potentials(MEPs)？ Dose individualized rTMS synchronized with motor training improve motor rehabilitation in patients without the ability to induce MEPs? Researchers will compare online rTMS to offline and sham stimulation in patients with MEPs to see if online rTMS works to alleviate motor dysfunction in preliminary trials. And compare individualized online rTMS to non-individualized online rTMS and sham in patients without MEPs to see if individualized online rTMS works to alleviate motor dysfunction in Randomized, double-blinded, and controlled trials.

Participants will:

randomized to one group acoording to the MEP condition of each person; receive rTMS treatment for 10 days, with 5 working days per week for a total of two weeks; receive magnetic resonance imaging (MRI) and electroencephalogram (EEG) evaluations before and after the entire treatment; conduct scales and MEP assessment one day before the treatment, as well as one day, one month, and three months after the treatment.

DETAILED DESCRIPTION:
In our experiment, patients were be randomly assigned to three groups: online, offline and sham groups. if patients were able to induce MEPs, intensity of TMS will be 80% RMT; if not , inensity of TMS will be 70% of TMS output.

ELIGIBILITY:
Inclusion Criteria:

1. The patient is first diagnosed with stroke through neurological examination, CT or MRI scan.
2. The vital signs are stable and there is a certain degree of upper limb motor dysfunction.
3. The age is between 20 and 80 years old.
4. The cognitive ability is not significantly affected and the patient can cooperate with various examinations and assessments, with a MMSE score ≥ 20 points.
5. There are no serious complications (such as pneumonia, heart failure, urinary tract infection or malnutrition).
6. There is no pathological condition that is a contraindication for TMS in the medical history (for example, patients with metal in the brain, such as aneurysm clips, patients with a cardiac pacemaker, pregnant women, or those with a history of epileptic seizures).
7. The patient or guardian agrees to sign the informed consent form.

Exclusion Criteria:

1. Patients with severe heart, lung, liver, kidney diseases and malignant tumors;
2. Those with a history of aphasia, severe cognitive impairment or mental illness;
3. Patients who have had a history of epileptic seizures in the last month or are taking anti-epileptic drugs recently;
4. Those with severe visual or hearing impairments, unable to communicate normally;
5. People with metal implants, pacemakers, skull defects or other conditions that prevent them from undergoing TMS.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-07-02 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Fugl-Meyer Assessment - Upper Extremity (FMA-UE) | Baseline; Day 1 After 2-week intervention; Day 30 after 2-week intervention; Day 60 after 2-week intervention
  The Fugl-Meyer Assessment (FMA) is a stroke-specific, performance-based impairment index. It is designed to assess motor functioning, balance, sensation and joint functioning in patients with post-stroke hemiplegia. It is applied clinically and in research to determine disease severity, describe motor recovery, and to plan and assess treatment.
  The Fugl-Meyer Assessment - Upper Extremity (FMA-UE) is the upper limb motor domain includes items assessing movement, coordination, and reflex action of the shoulder, elbow, forearm, wrist, hand. It ranges from 0 (hemiplegia) to 66 points (normal motor performance).

SECONDARY OUTCOMES:
Modified Barthel Index (MBI) | Baseline; Day 1 After 2-week intervention; Day 30 after 2-week intervention; Day 60 after 2-week intervention
  The Barthel Index for activities of daily living was introduced in 1965 by Barthel and Mahoney to be used in the assessment of the degree of assistance required by patients with stroke (other neuromuscular or musculoskeletal disorders or oncology patients) with regards to 10 items of mobility and self-care (ADL).
The Pittsburgh Sleep Quality Index (PSQI) | Baseline; Day 1 After 2-week intervention; Day 30 after 2-week intervention; Day 60 after 2-week intervention
  The Pittsburgh Sleep Quality Index (PSQI) is a widely used self-report questionnaire that assesses sleep quality over a one-month time interval.
  The PSQI is commonly used in both clinical and research settings to evaluate various aspects of sleep. It is a valuable tool for assessing sleep quality as it captures multiple dimensions of sleep, including both subjective experiences and objective parameters. It allows researchers and healthcare providers alike to obtain a comprehensive understanding of an individual's sleep patterns and disturbances and inform treatment decisions and interventions for sleep disorders.
Motor Evoked Potential (MEP) - Resting Motor Threshold (RMT) | Baseline; Day 1 After 2-week intervention; Day 30 after 2-week intervention; Day 60 after 2-week intervention
  Resting motor threshold is an objective measure of cortical excitability. Numerous studies indicate that the success of motor recovery after stroke is significantly determined by the direction and extent of cortical excitability changes.
The average completion time for baseline tasks | Day 1, Day 2, Day 3, Day 4, Day 5, Day 6, Day7, Day 8, Day 9, Day 10 during TMS intervention
  The average completion time for baseline tasks refers to the time (seconds) taken by the patient to complete the baseline motor task before each intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital of the Chinese People's Liberation Army Naval Medical University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
The investigators will share the demographic information and baseline clinical data of all participants.
Supporting Information: Study Protocol, SAP, CSR
Access Criteria: Authorized professional researchers, including but not limited to researchers engaged in neuroscience research who have obtained data access permission from their affiliated institutions, and clinical doctors from other medical institutions that have a cooperative relationship with this study and have signed data confidentiality agreements.
  They can access the detailed clinical medical histories of the participants, including past disease histories and treatment process records; neurological function assessment scale data; as well as imaging data collected during the study, such as brain magnetic resonance imaging (MRI) results. However, sensitive information related to participants' privacy, such as names, ID numbers, and contact information, will be strictly anonymized to ensure that such information cannot be obtained.
  They can contact the corresponding author or the first author via email.